CLINICAL TRIAL: NCT01817322
Title: Kidney Graft Function Under the Immunosuppression Strategies With Low Dose of Neoral®(Cyclosporine) and Standard Dose of Myfortic®(Enteric-Coated Mycophenolate Sodium) vs. With Conventional Dose of Neoral®(Cyclosporine) and Reduced Dose of Myfortic®(Enteric-Coated Mycophenolate Sodium) in De Novo Renal Transplant Recipients
Brief Title: Kidney Graft Function Under the Immunosuppression Strategies
Acronym: MyLowCsA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Joo Kim, Surgery M.D, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AKR09T
Record Dates: First submitted 2013-03-08; First posted 2013-03-25 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Renal Disease
Keywords: kidney transplantation
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Mycophenolic Acid; Prednisolone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myfortic® (Enteric-coated Mycophenolate Sodium) (Experimental): reduced cyclosporine+steroids+standard dose of myfortic
  Interventions: Drug: Standard Dose of Myfortic and Reduced Dose of Myfortic; Drug: Prednisolone OR methylprednisolone OR deflazacort injected both control group and experimental group; Drug: Basiliximab injected both control group and experimental group
- Myfortic (Active Comparator): Conventional Dose+cyclosporine+steroid+Reduced Dose of Myfortic
  Interventions: Drug: Standard Dose of Myfortic and Reduced Dose of Myfortic; Drug: Prednisolone OR methylprednisolone OR deflazacort injected both control group and experimental group; Drug: Basiliximab injected both control group and experimental group

INTERVENTIONS:
Drug: Standard Dose of Myfortic and Reduced Dose of Myfortic — Low Dose of Neoral (Cyclosporine) and Standard Dose of Myfortic (Enteric-Coated Mycophenolate Sodium) vs. with Conventional Dose of Neoral (Cyclosporine) and Reduced Dose of Myfortic (Enteric-Coated Mycophenolate Sodium)
  Other Names: Kidney Graft Function under the Immunosuppression Strategies
Drug: Prednisolone OR methylprednisolone OR deflazacort injected both control group and experimental group — 500 mg IV Injection in OP Day and 250 mg IV injection in POD1(1 Post op day). And then the drug dose is gradually reduced following the study institution's protocol. But the subject must be take the dose of 5mg of the drug per one day. The drug dose should be controlled on the basis of 5mg of Prednisolone. It can be used with the same dose of methylprednisolone 4 mg or deflazacort 6 mg.
  Other Names: Kidney Graft Function under the Immunosuppression Strategies
Drug: Basiliximab injected both control group and experimental group — The subject must be injected 20 mg of Simulect in Kidney transplantation day and just before the OP. After 4 days(96hour ± 12hr), the subject must be injected 20mg of Simulect, again.
  Other Names: Kidney Graft Function under the Immunosuppression Strategies

SUMMARY:
To demonstrate that cyclosporine-sparing immunosuppressions with the standard dose of Enteric-Coated Mycophenolate Sodium would preserve renal graft function after transplantation without an increase of incidences of adverse events, such as biopsy confirmed acute rejection, local or systemic infections, and bone marrow suppression.

DETAILED DESCRIPTION:
This clinical investigation will be the open-label, prospective, multi-center, 1:1 randomized comparative, longitudinal, and investigator-initiated study. Patients with end-stage renal disease will be assessed for the eligibility, and then be randomized using random number table into one of two groups prior to kidney transplantation.

Immunosuppression consisted of Cyclosporine(Neoral®), Methylprednisolone OR prednisone OR deflazacort(Brand name is not designated) and Enteric-Coated Mycophenolate Sodium(Myfortic®). Basilixumab(Simulect®) will be given just prior to transplant and 4 days after transplantation. The Enteric-Coated Mycophenolate Sodium will be given orally at the dose of 720 mg BID for Group A (investigational) or 360 mg BID for Group B (comparator), starting at two days after transplantation, as shown in the figure below. Cyclosporine will be given orally at a dose of 10 mg/Kg/day starting at a day before transplantation. Within a month after transplantation, the dose of the drug will be individually adjusted with goal trough blood level between 100 ng/mL and 200 ng/mL for Group A or between 200 ng/mL and 300 ng/mL for Group B, as displayed in the table below. From a month to 2 months post-transplantation, the target blood trough levels of cyclosporine will be reduced to between 75 ng/mL and 150 ng/mL for Group A or between 150 ng/mL and 250 ng/mL for Group B. From 2 months to 4 months post-transplantation, it will be further reduced to between 50 ng/mL and 125 ng/mL for Group A or between 125 ng/mL and 200 ng/mL for Group B. After 4 months post-transplantation, it will be further reduced to between 50 ng/mL and 100 ng/mL for Group A or between 100 ng/mL and 200 ng/mL for Group B.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with end-stage renal disease aged 20 to 65 years undergoing primary kidney transplantation
2. Kidney recipients who should be transplanted a kidney from a decease or living donor aged between 15 and 65 years
3. Patients who have given written informed consent to participate in the study

Exclusion Criteria:

* 1. multi-organ recipients, or dual kidney recipients or previous transplant recipients with any organs including the kidney ,bone marrow, or stem cells.

  2. Recipients who should be transplanted the kidney from a non-heart beating donor, an ABO incompatible donor ,or a lymphocyte cross-match positive donor 3. Patients with a history of malignancy within the last five years, except for successfully excised squamous or basal cell carcinoma of the skin.

  4. Patients with hypersensitivity to Mycophenolate sodium, Mycophenolate acid or Mycophenolate Mofetil or to any of the excipients.

  5. Patient with HGPRT(Hypoxanthin e-guanine phosphoribosyl-transferas) such as Lesch-Nyhan syndrome and kelley-Seegmiller syndrome.

  6. Patients who have tested positive for HIV, HCV and HBV surface antigen. 7. Recipients of organs from donors who tested positive for HBsAg, HCV, HIV 8. Patients with any known hypersensitivity to cyclosporine or other components of the formulations 9. Patients who are applicable to the contradiction of Sandimune Neoral 10. Patients who have received any investigational drug within 30 days prior to study entry.

  11. Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception.

  12. Existence of any surgical or medical condition, other than the current transplant, which in the opinion of the investigator might significantly alter the absorption, distribution, metabolism or excretion of study medication, and/or presence of severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus.

  13. Evidence of drug, alcohol abuse, and/or other psychiatric illness within the last 6 months prior to study enroll 14. At the time of the screen evaluation for this study, patients with platelet count<50,000/mm3, absolute neutrophil count of <1,500/mm3, white blood cell count of < 4,500/mm3, or patients who have an abnormal liver profile such as ALT, AST Alk Phos or total bilirubin>3 times the upper normal limit.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
eGFR (abbreviated MDRD equation) | 6 months after transplantation
  Primary objective: To compare the renal function with eGFR (abbreviated MDRD equation) 6 months after transplantation

SECONDARY OUTCOMES:
safety | 6 months after transplantation
  graft survival and patient survival

CONTACTS AND LOCATIONS:
Overall Officials: Jong won HA, M.D, Principal Investigator — Seoul National University Hospital; Myoung-soo kim, M.D, Principal Investigator — Yonsei University; chang-Kwon OH, M.D, Principal Investigator — Ajou unversity medical center